CLINICAL TRIAL: NCT04021368
Title: A Phase Ib Study of RVU120 (SEL120) in Patients With Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome
Brief Title: RVU120 in Patients With Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ryvu Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI120-001
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia; High-risk Myelodysplastic Syndrome
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndrome; CDK8/19 Inhibitor; RVU120 (SEL120); Clinical Trial, Phase Ib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Dose escalating Cohorts with a safety expansion Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RVU120(SEL120) (Experimental): The first part of the study consists of dose-escalation cohorts where patients will receive ascending doses of RVU120(SEL120) to determine the recommended dose (RD) for further clinical development. The second part of the study is an enrichment cohort where additional 6 to 20 patients will be treated with RVU120(SEL120) to support the evaluation of the RD.
  Interventions: Drug: RVU120(SEL120)

INTERVENTIONS:
Drug: RVU120(SEL120) — RVU120(SEL120) will be administered as a single oral dose every other day (q.o.d.) for a total of 7 doses i.e. on Days 1, 3, 5, 7, 9, 11 and 13, in a 3-week treatment cycle.

SUMMARY:
This first-in-human study will evaluate RVU120 (SEL120), a novel small molecule CDK8/19 inhibitor, in patients with Acute Myeloid Leukemia (AML) or High-risk Myelodysplastic Syndrome (HR-MDS), in terms of selection of the recommended dose for further clinical development and assessment of safety, tolerability, preliminary anti-leukemic activity, as well as pharmacokinetic and pharmacodynamic profiles.

DETAILED DESCRIPTION:
The study will determine the recommended phase II dose (RP2D) and safety of RVU120 (SEL120) given as monotherapy over a range of dose-levels, following a closely controlled dose escalation study design.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be met for a patient to be eligible for the study:

1. Written informed consent provided prior to any study-related procedure.
2. Age ≥18 years.
3. AML diagnosis according to the 2016 World Health Organisation (WHO) classification (Arber et al. 2016) with relapsed or refractory disease with no available therapy who have exhausted the applicable standard of care; or Myelodysplastic Syndrome (MDS) diagnosis according to the 2016 WHO classification (Arber et al. 2016) with high-risk disease per the Revised International Prognostic Scoring System (IPSS-R >4.5) and with relapsed or refractory disease with no available therapy who have exhausted the applicable standard of care.
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
5. Patients must have been off anti-cancer treatment prior to study.
6. Patients must have recovered from the toxic effects of previous treatments.
7. Peripheral white blood cell (WBC) count <10x10^9/L; Platelet count >10,000/μL; Serum albumin ≥ 30g/L (3.0g/dL); Normal coagulation (elevated INR, prothrombin time or APTT <1.3 x ULN acceptable); AST and ALT ≤3x ULN; Total bilirubin ≤1.5 x ULN; Creatinine clearance ≥60 mL/min (Cockcroft-Gault formula);
8. Adequate cardiac function
9. Life expectancy of at least 12 weeks.
10. For females of childbearing potential (FCBP), a negative pregnancy test must be confirmed before enrolment. FCBP must commit to use a highly effective method of contraception during study participation and until 6 months after the last dose of study drug. Females must also refrain from donating blood or egg (ovum) during the same time period.
11. For males, an effective barrier method of contraception must be used during study participation until 6 months after the last dose of study drug, if the patient is sexually active with a FCBP. Males must also refrain from donating blood or sperm during the same time-period.
12. Investigator considers the patient to be suitable for participation in the clinical study

Exclusion Criteria:

1. Active central nervous system (CNS) leukemia.
2. Previous treatment with CDK8-targeted therapy.
3. Patients who have undergone major surgery within 28 days prior to first dose of study drug.
4. Hematopoietic stem cell transplant within 120 days prior to first dose of study drug.
5. Active acute graft versus host disease (GVHD)
6. Infections and acute inflammatory conditions
7. Known seropositivity or history of HIV
8. Known positive test of / or known active diagnosis of COVID-19 viral infection
9. Ongoing significant liver disease
10. Impairment of gastrointestinal function or gastrointestinal disease
11. Ongoing drug-induced pneumonitis.
12. Concurrent participation in another investigational clinical trial.
13. Taking any medications, herbal supplements or other substances (including smoking) that are known to be strong inhibitors or inducers of CYP1A2 or that can prolong Q wave to T wave (QT) interval and/or cause torsade de pointes within less than 5 half-lives, prior to first dose of study drug.
14. Significant cardiac dysfunction or poorly controlled angina.
15. Currently taking drugs that are documented, in the drug package insert, to have a risk of causing prolonged QTc or torsades de pointes (TdP) within 5 half-lives prior to first dose of study drug.
16. Personal or family history of serious ventricular arrhythmia, or QT interval corrected for heart rate (QTc) ≥470 ms (Bazett's formula).
17. Any other prior or current medical condition or extenuating circumstance that, in the Investigator's opinion, could jeopardize patient safety or interfere with the objectives of the study.
18. Prior history of malignancies other than AML or MDS, unless the patient has been free of the disease for 5 years or more prior to Screening.
19. Pregnant or breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended dose (RD) | Up to 2 years
  The RD will be determined using all available data, which will include dose limiting toxicities (DLTs) and other toxicities, signs of anti-leukemic activity, pharmacokinetic and pharmacodynamic characteristics.
Incidence of Adverse Events (Safety and Tolerability) | Up to 2 years
  Safety and tolerability profile will be assessed by Common Terminology Criteria for Adverse Events v5.0 and summarized by type, frequency, and severity of adverse events.

SECONDARY OUTCOMES:
The Maximum Observed Concentration (C[max]) | Up to 2 years
  Pharmacokinetic profile of RVU120(SEL120) will be characterized using the Maximum Observed Concentration (C[max]).
The Terminal Half-life (t[1/2]) | Up to 2 years
  Pharmacokinetic profile of RVU120(SEL120) will be characterized using the Terminal Half-life (t[1/2]).
The Area Under the Curve (AUC) | Up to 2 years
  Pharmacokinetic profile of RVU120(SEL120) will be characterized using the Area Under the Curve (AUC).
The Volume of Distribution at Steady State (Vss) | Up to 2 years
  Pharmacokinetic profile of RVU120(SEL120) will be characterized using the Volume of Distribution at Steady State (Vss).
Anti-leukemic activity | Up to 2 years
  Anti-leukemic activity will be assessed by AML or MDS Response Criteria (Döhner et al., 2017, or Cheson et al., 2006, respectively).

OTHER OUTCOMES:
AML surface markers | Up to 2 years
  Pharmacodynamic profile of RVU120(SEL120) will be characterized using immunophenotyping of AML surface markers by exploratory assay.
Phosphorylated protein levels in AML blasts | Up to 2 years
  Pharmacodynamic profile of RVU120(SEL120) will be characterized using phosphorylated protein levels in AML blasts by exploratory immunoassay.
Transcriptomic profile changes in AML blasts | Up to 2 years
  Pharmacodynamic profile of RVU120(SEL120) will be characterized using transcriptomic profile changes in AML blasts by exploratory next generation sequencing.
Genetic profile changes in AML blasts | Up to 2 years
  Pharmacodynamic profile of RVU120(SEL120) will be characterized using genetic profile changes in AML blasts by next generation sequencing.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (5):
  - Sylvester Comprehensive Cancer Center, University of Miami Hospital and Clinics, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - MICS Centrum Medyczne Toruń, Torun
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Dolnośląskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
  - Świętokrzyskie Centrum Onkologii, Klinika Hematologii i Transplantacji Szpiku, Kielce, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: No